CLINICAL TRIAL: NCT05021367
Title: A Phase I Clinical Trial to Evaluate the Safety and Tolerability of TQB3823 Tablets in Subjects With Advanced Malignancies
Brief Title: A Clinical Study of TQB3823 in Patients With Advanced Malignant Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3823-I-01
Record Dates: First submitted 2021-08-24; First posted 2021-08-25 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3823 tablets (Experimental): Subjects receive TQB3823 in the first cycle for a total of 28 days , a single dose on Day 1. Day 2 to Day 7 are the elution period, and the continuous doses are from Day 8 to Day 21. From the second cycle, continuous treatment for 28 days is as a treatment cycle.
  Interventions: Drug: TQB3823 tablets

INTERVENTIONS:
Drug: TQB3823 tablets — TQB3823 is a small molecule Poly ADP-ribose Polymerase (PARP) inhibitor that can inhibit the enzyme activity of PARP1/2, making it difficult to repair the DNA in cancer cells, leading to cell death and delaying or blocking tumor development.

SUMMARY:
This is a study to evaluate the maximum tolerated dose (MTD) , occurrence of all adverse events (AEs) and serious adverse events (SAEs) , pharmacokinetic parameters and antitumor effect of TQB3823 tablets in Chinese adult patients with advanced solid tumors .The study was divided into phase Ia and phase Ib, Phase Ia: Dose escalation period, to evaluate the safety and tolerability of TQB3823 tablets, determine MTD;Phase Ib: Effectiveness exploration period, to expand the safe and effective dose group, and to recommend appropriate dosage and method for subsequent clinical research.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily join the study, sign the informed consent form, and have good compliance.
2. Aged from 18 to 75 years; Eastern Cooperative Oncology Group (ECOG) performance status score: 0-1; at least 3 months expected survival period.
3. Subjects with relapse advanced malignant solid tumors clearly diagnosed by pathology and / or cytology, lack of conventional effective treatment methods.
4. The function of main organs is normal.
5. Subjects need to adopt effective methods of contraception.

Exclusion Criteria:

1. Subjects with other malignancies currently or suffered within 3 years. The following two conditions can be enrolled: other malignant tumors treated with a single operation to achieve disease-free survival (DFS) for 5 consecutive years; cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors[ Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)].
2. Subjects with multiple factors affecting oral administration.
3. Subjets with unhealed toxicity above Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 due to previous antitumor treatment.
4. Subjects who have received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before first administration.
5. Subjects with long lasting wounds or fractures.
6. Subjects with a history of psychotropic drug abuse unable to quit or with mental disorders.
7. Subjects with any severe and/or uncontrolled disease.
8. Subjects who have received surgery, chemotherapy, radiotherapy or other anticancer therapies 4 weeks before the first administration ( 2 weeks for brain radiotherapy ).
9. Subjects who have taken Chinese patent medicines with anti-tumor indications in the drug instructions that National Medical Products Administration (NMPA)approved within 2 weeks before the first administration.
10. Subjects with pleural effusion, pericardial effusion or ascites that cannot be controlled and need repeated drainage.
11. Subjects with known central nervous system metastases and/or cancerous meningitis.
12. Subjects who have participated in other clinical studies within 4 weeks before the first administration.
13. According to the judgment of the investigators, there are accompanying diseases that seriously endanger the safety of patients or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Baseline up to 28 days
  Subjects within 28 days after treatment appear the following toxicity reaction relate to the drug ：III °or above of non-hematological toxicity, IV°hematological toxicity ,Neutropenia associated with fever.
Maximum tolerated dose (MTD) | Baseline up to 28 days
  The highest dose at which no more than 33% of the subjects experience a dose-limiting toxicity (DLT) during treatment

SECONDARY OUTCOMES:
Adverse events (AEs) and serious adverse events (SAEs) | Baseline up to 28 days
  The occurrence of all AEs and SAEs，such as Anemia, Platelet count decreased, Nausea, Vomiting, Elevated transaminase.
Overall response rate (ORR) | 21 days
  Overall response rate（From the first drug treatment to the last drug treatment）
Disease control rate（DCR） | 21 days
  Disease control rate（From the first drug treatment to the last drug treatment）
Progression-free survival (PFS) | 21 days
  First-time progression of disease/ recurrence /death）
Duration of Response (DOR) | 21 days
  Baseline up to progression of disease/ recurrence /death
Time to reach maximum (peak) plasma concentration following drug administration（Tmax） | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  To characterize the pharmacokinetics of TQB3823 by assessment of time to reach maximum plasma concentration after single and multiple dosing
Maximum (peak) plasma drug concentration （Cmax） | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  Cmax is the maximum plasma concentration of TQB3823 or metabolite(s).
Maximum (peak) steady-state plasma drug concentration during a dosage interval （Cmax,ss） | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  Cmax is the maximum plasma concentration of TQB3823 or metabolite(s).
Area under the plasma concentration-time curve from time zero to time t （AUC0-t）、Area under the plasma concentration-time curve from time zero to infinity （ACU0-∞） | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  To characterize the pharmacokinetics of TQB3823 by assessment of area under the plasma concentration time curve from the first dose to infinity.
Apparent total clearance of the drug from plasma after oral administration （CL/f） | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  CL/f is total clearance rate for TQB3823.
Elimination half-life（t1/2） | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  t1/2 is time it takes for the blood concentration of TQB3823 or metabolite(s) to drop by half.
Mean residence time (MRT) | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  MRT describes the average time that TQB3823 or metabolite(s) remain in the body.
Minimum steady-state plasma drug concentration during a dosage interval （Css-min） | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  Css-min is the minimum plasma concentration of TQB3823 or metabolite(s).
Average steady-state plasma drug concentration during multiple-dose administration （Css-av） | Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24, 48, 72, 120, 168 hours post-dose on single dose; Hour 0(pre-dose) of day 7,day 14 on multiple dose and Hour 0 (pre-dose), 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on multiple dose of day 21.
  Css-av is mean steady-state plasma concentration of TQB3823 or metabolite(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Cen, Guangzhou, Guangdong, China